CLINICAL TRIAL: NCT02467712
Title: Change in Joint Prosthesis in One Step Due to Fungal Infection
Brief Title: Fungal Infection on a Joint Prosthesis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 2014-67
Record Dates: First submitted 2015-06-07; First posted 2015-06-10 (Estimated); Last update posted 2015-06-10 (Estimated); Status verified 2015-06

CONDITIONS: Fongal Infection
Keywords: Fongal infection; joint prosthesis; prosthetic reconstruction

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
It is generally accepted that the fungal infection on a joint prosthesis is to be treated in two surgical time: implant removal and prosthetic reconstruction. The service took the option for over 10 years to treat bacterial infections in joint replacement by a change in time. In four recent cases the diagnosis initially suspected of bacterial infection has been restated on intraoperative bacteriological examinations fungal infection. It is therefore a potentially harmful side effect of the chosen treatment option, but 4 patients in question were all cured of their fungal infection after a postoperative antifungal therapy. The objective of this study is to report these cases for discussion on the therapeutic choices in fungal infections on joint replacement.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years
* Patient having surgery for the management of fungal infection after change in one step in joint replacement prothesis in the participating services in 2014.

Exclusion Criteria:

* Patients under 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients over 18 years having surgery for the management of fungal infection after change in one step in joint replacement prothesis in the participating services in 2014.
Sampling Method: Non-Probability Sample
Enrollment: 4 (Estimated)
Dates: Start 2015-07; Primary Completion 2016-07 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
Fungal infection | for the duration of hospital stay, up to 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Yves JENNY, MD, Principal Investigator — University Hospital, Strasbourg, France